CLINICAL TRIAL: NCT03006757
Title: Measurement of the Biting Force of Rabid Heat Cured Acrylic Resin Versus Modified Conventional Acrylic Resin With Titanium Dioxide Nanoparticles in Maxillary Single Dentures
Brief Title: Measurement of the Biting Force of Rabid Heat Cured Acrylic Resin Versus Modified Conventional Acrylic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: emad gamal ismail (Other)
Responsible Party: Sponsor-Investigator, emad gamal ismail, principal invistigator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 900
Record Dates: First submitted 2016-12-16; First posted 2016-12-30 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Column titanium dioxide (Experimental): patient take titanium dioxide denture participants will receive titanium dioxide denture ( made from conventional acrylic resin modified by titanium dioxide nanoparticles ) for 1 month in the initial phase of the trial.
  Interventions: Other: titanium dioxide denture base
- column placebo (Experimental): patient will take denture with conventional acrylic ( 20 minutes cure ) for 1 month in the initial phase
  Interventions: Other: titanium dioxide denture base

INTERVENTIONS:
Other: titanium dioxide denture base

SUMMARY:
The purpose of this study is to compare the effect of rapid heat cured acrylic resin material with titanium dioxide nanoparticles added to conventional acrylic resin material on the biting force of the single maxillary complete denture .

DETAILED DESCRIPTION:
Bite force is one indicator of the functional state of the masticatory system that results from the action of jaw elevator muscles modified by the craniomandibular biomechanics .Determination of individual bite force level has been widely used in dentistry, mainly to understand the mechanics of mastication for evaluation of the therapeutic effects of prosthetic devices and to provide reference values for studies on the biomechanics of prosthetic devices. In addition, bite force has been considered important in the diagnosis of the disturbances of the stomatognathic system .

Twenty (20) single maxillary completely edentulous patients were selected from the out-patient clinic of the Removable Prosthodontics Department, Faculty of Oral and Dental Medicine, Cairo University.

The primary outcome is to measure the biting force of single maxillary complete denture by I Load star sensor .

ELIGIBILITY:
Inclusion Criteria:

* completely edentulous maxillary arch and full or partial dentate mandibular arch with adequate inter arch space
* edentuluos arches should be covered by firm healthy mucosa angle class 1 maxillomandibular relationship

Exclusion Criteria:

* patients with bad habits
* previous history of radiotherapy or chemotherapy

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
measurement of the biting force of rabid heat cured acrylic resin versus modified conventional acrylic with titanium dioxide nanoparticles in maxillary single denture using i load star sensor | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mahmoud Adly, Giza, Giza Governorate, Egypt